CLINICAL TRIAL: NCT01127997
Title: The Effect and Mechanisms of the Second-meal Phenomenon in Type 2 Diabetic
Brief Title: The Effect and Mechanisms of the Second-meal Phenomenon in Type 2 Diabetic Patients
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Seung-Hwan Lee, The Catholic University of Korea
Other Study IDs: VC10EISI0007
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2010-08-23 (Estimated); Status verified 2010-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- study A: post-breakfast meal tolerance test + post-lunch meal tolerance test
- study B: fasting + post-lunch meal tolerance test

SUMMARY:
Second-meal phenomenon denotes the effect of a prior meal in decreasing the rise in blood glucose after a subsequent meal. This phenomenon occurs in normal subjects while it is not clear whether it is also observed in type 2 diabetic patients. This study aims to define whether the second-meal phenomenon occurs in type 2 diabetic patients. We will also seek for the mechanism.

ELIGIBILITY:
Inclusion Criteria:

* age 35-70
* HbA1c 6-8%
* DM duration less than 5 yrs

Exclusion Criteria:

* type 1 DM, secondary DM, gestational DM
* patients using insulin, TZDs
* patients using corticosteroid, herb medication or other medications affecting glucose tolerance
* renal dysfunction (Cr > 1.5mg/dL)
* hepatic dysfunction (LFT > x 3UNL)
* anemia (Hg < 10g/dL)
* ischemic heart disease, congestive heart failure
* severe diabetic complication (CRF, CVA, PDR, gastroparesis)
* infectious disease
* malignancy
* pregnant women

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type 2 diabetic patients
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Area under the curve of plasma glucose after meal | 3 months
  Compare the post-lunch AUC of glucose between two meal tolerance tests(one after having breakfast, one after not having breakfast)

SECONDARY OUTCOMES:
the mechanism of second-meal phenomenon | 3 months
  serum FFA, plasma insulin, C-peptide, incretin concentration will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- St. Vincent's hospital, Suwon, Kyounggi-do, South Korea

REFERENCES:
- [Background] Jovanovic A, Leverton E, Solanky B, Ravikumar B, Snaar JE, Morris PG, Taylor R. The second-meal phenomenon is associated with enhanced muscle glycogen storage in humans. Clin Sci (Lond). 2009 Jul 2;117(3):119-27. doi: 10.1042/CS20080542. PMID 19161346
- [Background] Bonuccelli S, Muscelli E, Gastaldelli A, Barsotti E, Astiarraga BD, Holst JJ, Mari A, Ferrannini E. Improved tolerance to sequential glucose loading (Staub-Traugott effect): size and mechanisms. Am J Physiol Endocrinol Metab. 2009 Aug;297(2):E532-7. doi: 10.1152/ajpendo.00127.2009. Epub 2009 Jun 16. PMID 19531643
- [Result] Jovanovic A, Gerrard J, Taylor R. The second-meal phenomenon in type 2 diabetes. Diabetes Care. 2009 Jul;32(7):1199-201. doi: 10.2337/dc08-2196. Epub 2009 Apr 14. PMID 19366973
- [Derived] Lee SH, Tura A, Mari A, Ko SH, Kwon HS, Song KH, Yoon KH, Lee KW, Ahn YB. Potentiation of the early-phase insulin response by a prior meal contributes to the second-meal phenomenon in type 2 diabetes. Am J Physiol Endocrinol Metab. 2011 Nov;301(5):E984-90. doi: 10.1152/ajpendo.00244.2011. Epub 2011 Aug 9. PMID 21828339